CLINICAL TRIAL: NCT05622435
Title: Clinical Investigation to Evaluate the Tolerance of T10070 on Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LT10070-001
Record Dates: First submitted 2022-10-12; First posted 2022-11-18 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T10070 (Experimental)
  Interventions: Device: T10070, Plastic tube with a roll-on applicator filled with an ointment

INTERVENTIONS:
Device: T10070, Plastic tube with a roll-on applicator filled with an ointment — 6 times per day on both (upper and lower) eyelids of right eye during 7 to 9 days.

SUMMARY:
The goal of this clinical trial investigation is to evaluate the tolerance of the T10070 on healthy volunteers by clinical examination under ophthalmological control.

Participants will attend 2 visits (inclusion at day 0 and follow-up/final at D7/D9. After inclusion, subjects will have to apply T10070 6 times a day during 7 to 9 days. The following tasks will be asked to participants:

* ophtalmological examination
* diary completion to record T10070 applications, potential discomfort/reactions observed and medication taken.
* complete subject questionnaire about usability of the product

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated
* Subject ≥ 18 years old
* Healthy volunteer
* Normal ocular examination in both eyes
* Normal skin examination in both eyes

Main Exclusion Criteria:

* Far best-corrected visual acuity (BCVA) ≥ +0.1 LogMar (e.g., ≤ 0.8 in decimal value or ≤ 80/100 Snellen equivalent)
* Known or suspected hypersensitivity to one of the components of the T10070
* History of trauma, infection, clinically significant inflammation within the 3 previous months
* Ongoing or know history of ocular allergy and/or uveitis and/or viral infection
* Diagnosed keratoconus
* Any palpebral abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in clinical examination on eyes and peri-ocular skin | signs assessment at Day 0 and Day 7/Day 9
  A clinical examination will be performed before and after product use on eyes and peri-ocular skin using 5-point structured scales (from "Absence (0)" to "Severe (4)") to evaluate the intensity of several signs.
Change from baseline in subjective evaluation of ocular and cutaneous signs by subjects | Signs assessment at Day 0 and Day 7/Day 9
  A subjective tolerance evaluation will be performed before and after product use using 5-point structured scales (from "No reaction (0)" to "Severe (4)").
Local tolerance assessed by Investigator | Local tolerance assessed at Day 7/Day 9
  Assessed using a 4-point scale (from "Bad tolerance" to "Very good tolerance").

SECONDARY OUTCOMES:
Subject questionnaire on product usability | Day 7/Day 9
  The subjective evaluation of the tested medical device will be assessed by subject by answering a satisfaction questionnaire. For each question, there are 4 possible answers (agree, somewhat agree, somewhat disagree, disagree)
Adverse Events | Day 7/Day 9
  Proportion of subjects experiencing at least one AE/SAE, TEAE related to the device, Serious TEAE.

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Paw, Doctor, Principal Investigator — Eurofins Dermscan Poland
Locations (1):
- Eurofins Dermscan Poland, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No